CLINICAL TRIAL: NCT02696733
Title: Ultrasound-Guided Obturator Nerve Block for Transurethral Procedures - Interadductor Approach
Brief Title: Ultrasound-Guided ONB for Transurethral Procedures - Interadductor Approach
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Karolina Dobrońska, M.D., Medical University of Warsaw
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U/1/2014
Record Dates: First submitted 2016-02-22; First posted 2016-03-02 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Urinary Bladder Neoplasms; Transurethral Resection; Nerve Block
Keywords: TURBT; ultrasound guided; ONB; interadductor approach
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UG - ONB (Experimental): Patients with the bladder tumor located on the lateral wall, with the high risk of adductor muscles contraction during TURBT under spinal anesthesia.
  Interventions: Device: Ultrasound; Drug: lidocaine 2%; Drug: 0.9% Natrium Chloratum with a 2nd generation cephalosporin

INTERVENTIONS:
Device: Ultrasound — Ultrasound-guided obturator nerve localization
  Other Names: USG
Drug: lidocaine 2% — local anesthetic used to block the obturator nerve
Drug: 0.9% Natrium Chloratum with a 2nd generation cephalosporin

SUMMARY:
Obturator nerve block is an effective method to prevent adductor muscles contraction during transurethral resection of bladder tumour localized on the lateral wall. Due to prior spinal anaesthesia the patient does not feel uncomfortable during the blockade and the interadductor approach gives the possibility to perform it in the lithotomy position. The aim of the study was to evaluate the safety and effectiveness of ultrasound-guided obturator nerve identification and blockade for TURBT.

DETAILED DESCRIPTION:
The basic methods for diagnosis and management of bladder cancer are endoscopic procedures. Transurethral resection of bladder tumor (TURBT) is usually performed under spinal anesthesia that does not prevent an unintended stimulation of the obturator nerve (ON) when electroresection is performed on the lateral wall of the bladder. This sensorimotor nerve arises from the lumbar plexus at L2-L4. It innervates the muscles responsible for adducting the thigh and the skin on the surface of the paramedian segment of the thigh. During TURBT, when the bladder has been filled with irrigation fluid, the ON is directly adjacent to the lateral wall of the bladder and it can be stimulated during the electroresection. Sudden contraction of the adductor muscles of the thigh, may lead to perforation of bladder wall with the resectoscope loop.

In the Department of General, Oncologic and Functional Urology, Medical University of Warsaw approximately 500 TURBT are performed every year; 7% of them necessitate the prevention of ON stimulation. Anesthetists perform obturator nerve block (ONB) - the anterior branch, using the stimulator for the identification with the 94% efficacy.

Recently, ultrasound guidance has been used to enhance the safety and efficacy of the nerve blocks that is why we have decided to evaluate the effectiveness of ONB performed with ultrasounds.

An approval from the Medical University of Warsaw Bioethical Committee has been obtained. Patients need to give written informed consent to participate in the study.

It is anticipated that 100 patients with TURBT performed under spinal anesthesia that, after the urologist decision, necessitate the ONB will be enrolled in this study.

Before the procedure an oral premedication is given. After admission to the operating room, intravenous access is established and the patient receives a drip infusion of 500 ml 0.9% Natrium Chloratum with an antibiotic (2nd generation cephalosporin). Constant monitoring is ensured of ECG, heart rate, and pulse oxymetry. Non-invasive blood pressure measurement is taken every five minutes. To maintain patients' blood oxygenation, oxygen is delivered with the use of a facemask. Spinal anesthesia is performed with patients in the sitting position, most frequently in the L3 L4 space (in the case of technical difficulties - L2 L3 or L4 L5) using 8-15 mg 0.5% hyperbaric bupivacaine depending on the patient's anthropometric parameters. The needles used are 25-27G pencil point. After drug administration, the patient is placed in the supine position.

Upon reaching the appropriate anesthesia level (Th10), which blocks conduction in the sensory nerve fibers of the bladder, the patient is placed in the lithotomy position. In the case of tumors located on the lateral wall of the bladder, the safety of TURBT is ensured using a neurotest performed by an urologist with a nerve stimulator built into the resectoscope (Neurotester FB2, ERBE). The extremity movement leads to the decision to block the ON.

Ultrasound-guided ONB procedure:

The patient remains in the lithotomy position. For nerve identification a linear transducer is used. It is placed next to the grain to visualize three adductor muscles. Between adductor longus and adductor brevis, in fascial plane, an anterior branch of obturator should be visualized. The needle is advanced toward the nerve in an out-of-plane trajectory. The local anesthetic is injected after heme-negative aspiration. The resistance during injection is avoided to reduce the risk of intraneural injection. If there are problems with nerve identification the anesthetic is injected in fascial plane between adductors muscles - longus and brevis.

10 ml of 2% lidocaine is used for single block and 2 x 10 ml of 2% lidocaine with epinephrine when bilateral one is needed.

Before TURBT starts again, the urologist once more perform the neurotest to evaluate the ONB efficacy.

After enrolling 50 patients to the study the results will be evaluated and the decision whether to decrease the amount of 10 ml of 2% lidocaine for injection will be taken.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* bladder tumor located on the lateral wall
* transurethral resection of the bladder tumor
* urologist decision that there is a risk of the stimulation of obturator nerve during resection
* spinal anesthesia

Exclusion Criteria:

* patients' refusal
* contraindications for spinal anesthesia
* skin lesions at injection site
* patients who really did not need ONB.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of ultrasound guided obturator nerve block - evaluated by a number of participants having transurethral resection of bladder tumor without unintended obturator nerve stimulation. | 30 months
  The investigator evaluates whether the urologist was able to perform safe electroresection of bladder tumor with no extremity movement. All extremity movements due to obturator nerve stimulation and all necessities to perform general anesthesia will be counted as unsuccessful ultrasound - guided ONB.

SECONDARY OUTCOMES:
Success rate of obturator nerve visualization with ultrasounds | 30 months
  The investigators evaluate whether it was possible to visualize the obturator nerve in the fascial plane
Efficacy of ONB - measured with nerve stimulator built in the resectoscope | 30 months
  A nerve stimulator (Neurotester FB2, ERBE) is used to evaluate the efficacy of the nerve block. Current flow settings are progressively marked relative to a 1-5 scale .
Safety of ultrasound-guided ONB measured by number of complications | 30 months
  hematoma , lidocaine overdose symptoms, bladder perforation,obturator nerve injury

CONTACTS AND LOCATIONS:
Overall Officials: Karolina Dobronska, MD, Principal Investigator — I Department of Anaesthesiology and Intensive Care
Locations (2):
- Poland (2):
  - I Department od Anaesthesiology and Intensive Care, Warsaw
  - I Department of Anaesthesiology and Intensive Care, Medical University of Warsaw, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pladzyk K, Jureczko L, Lazowski T. Over 500 obturator nerve blocks in the lithotomy position during transurethral resection of bladder tumor. Cent European J Urol. 2012;65(2):67-70. doi: 10.5173/ceju.2012.02.art2. Epub 2012 Jun 12. PMID 24578931
- [Result] Thallaj A, Rabah D. Efficacy of ultrasound-guided obturator nerve block in transurethral surgery. Saudi J Anaesth. 2011 Jan;5(1):42-4. doi: 10.4103/1658-354X.76507. PMID 21655015